CLINICAL TRIAL: NCT01419249
Title: First Year Growth Response Associated Genetic Markers Validation Phase IV Open-label Study in Growth Hormone Deficient and Turner Syndrome Pre-pubertal Children: the PREDICT Pharmacogenetics Validation Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck KGaA, Darmstadt, Germany (Industry)
Collaborators: Merck Serono S.A., Geneva (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: EMR 200104_010
Record Dates: First submitted 2011-08-16; First posted 2011-08-18 (Estimated); Results first posted 2014-01-16 (Estimated); Last update posted 2014-01-16 (Estimated); Status verified 2013-11

CONDITIONS: Idiopathic Growth Hormone Deficiency; Turner Syndrome
Keywords: Growth Hormone Deficiency; Turner syndrome; Pharmacogenetics; Recombinant Human Growth Hormone therapy
MeSH Terms: conditions — Turner Syndrome; Dwarfism, Pituitary | interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Retrospective cohort (Other)
  Interventions: Other: Blood sampling

INTERVENTIONS:
Other: Blood sampling — Subjects with pre-established diagnosis of IGHD and TS and were treated with r-hGH therapy for 1 year, will be observed in this retrospective cohort study wherein blood sampling will performed for genotyping of the various genetic markers along with collection of retrospective data relative to the r-hGH treatment.

SUMMARY:
PREDICT Validation is a validation pharmacogenetic trial. The purpose of this study is to confirm that some genes can be used to predict how well a subject diagnosed with idiopathic growth hormone deficiency (IGHD) or turner syndrome (TS) will respond to a treatment with recombinant human growth hormone (r-hGH).

DETAILED DESCRIPTION:
This study is an open-label, interventional, retrospective, multicenter, international study, single-arm, non-randomized, and non-controlled study. The subject's trial participation includes a single visit. During the visit, subjects who give consent to participate in the trial will undergo blood sampling for genetic markers testing and retrospective data will be collected relative to the first year of the subject's r-hGH treatment.

The r-hGH treatment followed by the subject is indicated the pediatric population, therefore most of the subjects included into the trial will be below 18 years old.

This study is a non-investigational medicinal product (IMP) trial therefore no drug product data is provided.

ELIGIBILITY:
Inclusion Criteria:

* Pre-established diagnosis of IGHD or TS based on classical criteria with at least 1 year of r-hGH therapy and with Tanner stage 1 at treatment start
* Retrospective availability of a complete set of clinical, auxological and biological parameters necessary for building the predictive model
* Other protocol defined inclusion criteria could apply

Exclusion Criteria:

* Acquired growth hormone deficiency (GHD)
* Any drug or disease that could affect growth during the first year of r-hGH treatment
* Other protocol defined exclusion criteria could apply

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 458 (Actual)
Dates: Start 2011-09; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Della Corte, Study Director — Merck Serono S.A. , Geneva, Switzerland
Locations (31):
- Argentina (3):
  - Hospital de Niños Ricardo Gutiérrez, Buenos Aires
  - Hospital de Pediatria Garrahan, Buenos Aires
  - Hospital de Niños de la Santisima Trinidad, Córdoba
- Canada (4):
  - University of Calgary - Alberta Children's Hospital, Calgary
  - CHU Sainte Justine Montréal, Montreal
  - Centre Hospitalier Universitaire de Sherbrooke - Fleurimont, Sherbrooke
  - British Columbia Children's Hospital, Vancouver
- Czechia (4):
  - Fakultní nemocnice Brno, Brno
  - University Hospital Hradec Kralove, Hradec Králové
  - Faculty Hospital, Olomouc
  - University Hospital Praha Motol, Prague
- France (3):
  - Centre d'Endocrinologie Pédiatrique, Bordeaux
  - CHU Bordeaux - Hopital pédiatrique Pellegrin, Bordeaux
  - Hôpital Femme-Mère-Enfant, Bron
- Germany (2):
  - University of Cologne Children's Hospital, Cologne
  - University Children's Hospital, München
- Italy (4):
  - University of Bari Aldo Moro, Bari
  - Ospedale Microcitemico di Cagliari, Cagliari
  - Centro di Endocrinologia e Diabetologia Pediatrica, Catania
  - Istituto Giannina Gaslini - Clinica Pediatrica, Genova
- Spain (5):
  - Hospital 12 de Octubre, Madrid
  - Hospital Infantil Universitario Niño Jesús, Madrid
  - Hospital Universitario Gregorio Maran, Madrid
  - Hospital Clínico Universitario de Santiago de Compostela, Santiago de Compostela
  - Hospital Miguel Servet, Zaragoza
- Sweden (3):
  - Queen Silvia Children's Hospital, Gothenburg
  - Faculty of Health Sciences, Linkping University, Linköping
  - Karolinska University Hospital Campus Solna, Stockholm
- United Kingdom (3):
  - Birmingham Children's Hospital, Birmingham
  - Royal Manchester Children's Hospital, Manchester
  - Sheffield Children's Hospital, Sheffield

RESULTS

PARTICIPANT FLOW:
Groups:
- Idiopathic Growth Hormone Deficiency (IGHD) Cohort: Participants with pre-established diagnosis of IGHD and were treated with recombinant human growth hormone (r-hGH) therapy for at least 1 year were observed in this retrospective cohort study wherein blood sampling was performed for genotyping of the various genetic markers along with collection of retrospective data relative to the r-hGH treatment.
- Turner Syndrome (TS) Cohort: Participants with pre-established diagnosis of TS and were treated with r-hGH therapy for at least 1 year were observed in this retrospective cohort study wherein blood sampling was performed for genotyping of the various genetic markers along with collection of retrospective data relative to the r-hGH treatment.
Period: Overall Study
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort
Started | 318 | 140
Completed | 318 | 140
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS) population included all the participants who had provided informed consent and had non-missing height at start (defined as within one month prior to treatment start date) and at 1 year (+/- 120 days) of r-hGH treatment and had pharmacogenomics data available.
Groups:
- Total: Total of all reporting groups
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort | Total
Number analyzed (Participants) | 293 | 132 | 425
Age, Customized [Number; unit: participants]
  less than (<) 8 years | 197 | 95 | 292
  Between 8 to 12 years | 84 | 31 | 115
  greater than (>) 12 years | 12 | 6 | 18
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 85 | 132 | 217
  Male | 208 | 0 | 208

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Height at Year 1
Description: Change from baseline in height at year 1 was one of the growth parameter to assess the first year growth response to r-hGH treatment.
Time Frame: Baseline and Year 1
Population: FAS population included all the participants who had provided informed consent and had non-missing height at start (defined as within one month prior to treatment start date) and at 1 year (+/- 120 days) of r-hGH treatment and had pharmacogenomics data available.
Measure: Mean (Standard Deviation); unit: centimeter
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort
Number analyzed (Participants) | 293 | 132
centimeter
  Baseline | 103.6 (18.1) | 103.5 (16.3)
  Change at Year 1 | 9.8 (2.7) | 8.6 (2.0)

2. Secondary Outcome: Evaluation of the Contribution of Validated Genetic Markers to the Amplitude of First Year Growth Response to r-hGH Therapy in IGHD Children Using Growth Hormone Deficiency Kabi-Pharmacia International Growth Study (GHD KIGS) Predictive Model
Description: GHD KIGS predictive model includes various clinical, auxological and biological markers which are as follows: maximum growth hormone (GH) response to provocation test; age at onset of therapy; birth weight SDS; average GH dose received during the first year of r-hGH therapy; height SDS at start of therapy; the difference between the pre-treatment height SDS of the subject and the mid parental height SDS; and weight SDS at start of therapy.
Time Frame: Year 1
Population: No genetic markers were identified during the study therefore, the data for this outcome measure was not analyzed.
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort
Number analyzed (Participants) | 0

3. Secondary Outcome: Evaluation of the Contribution of Validated Genetic Markers to the Amplitude of First Year Growth Response to r-hGH Therapy in TS Girls Using Turner Syndrome Kabi-Pharmacia International Growth Study (TS KIGS) Predictive Model
Description: TS KIGS predictive model includes various clinical, auxological and biological markers which are as follows: maximum GH response to provocation test; age at onset of therapy; birth weight SDS; average GH dose received during the first year of r-hGH therapy; height SDS at start of therapy; the difference between the pre-treatment height SDS of the subject and the mid parental height SDS; and weight SDS at start of therapy.
Time Frame: Year 1
Population: No genetic markers were identified during the study therefore, the data for this outcome measure was not analyzed.
Arm/Group | Turner Syndrome (TS) Cohort
Number analyzed (Participants) | 0

4. Primary Outcome: Change From Baseline in Height Standard Deviation Score (SDS) at Year 1
Description: Height SDS was calculated as height minus reference mean height divided by standard deviation of the reference population. Height SDS reflects the height relative to a reference population of the same age and gender. Change from baseline in height SDS at Year 1 was one of the growth parameter to assess the first year growth response to r-hGH treatment.
Time Frame: Baseline and Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort
Number analyzed (Participants) | 293 | 132
standard deviation score
  Baseline | -2.60 (1.06) | -2.17 (1.03)
  Change at Year 1 | 0.98 (0.67) | 0.71 (0.48)

5. Primary Outcome: Height Velocity Standard Deviation Score (SDS) at Year 1
Description: Height velocity SDS was calculated as height velocity minus reference mean height velocity divided by standard deviation of the reference population. Height velocity SDS reflects the height velocity relative to a reference population of the same age and gender. Height velocity SDS at Year 1 was one of the growth parameter to assess the first year growth response to r-hGH treatment.
Time Frame: Year 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: standard deviation score
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort
Number analyzed (Participants) | 293 | 132
standard deviation score | 4.18 (2.90) | 2.59 (1.92)

ADVERSE EVENTS:
Description: As it is a retrospective study, only serious adverse events which were considered by the investigator to be at least possibly related to the conduct of the trial were collected.
Arm/Group | Idiopathic Growth Hormone Deficiency (IGHD) Cohort | Turner Syndrome (TS) Cohort
Serious Adverse Events (participants affected / at risk) | 0/293 | 0/132
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
No genetic markers were identified, therefore data for the secondary outcome measures was not analyzed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor does not object to trial results publication by Investigator. Investigator will provide sponsor proposed publication/disclosure for review before submission. In multi-center trial, Investigator agree on first publication to be joint involving all sites. Investigator can decline to be part of joint publication. If joint manuscript has not submitted for publication within 12 months of trial completion/termination at all sites, Investigator can publish separately, subject to this agreement.